CLINICAL TRIAL: NCT02958410
Title: A Clinical Research of CD30-Targeted CAR-T in Lymphocyte Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Shiqi Li, Principal Investigator of Biotherapy Center, Southwest Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMMU-BTC-010
Record Dates: First submitted 2016-11-06; First posted 2016-11-08 (Estimated); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Leukemia; Lymphoma
Keywords: CD30; CAR-T
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lymphocyte Malignancies (Experimental): The trial will be conducted in a manner of simon two-stage design with Anti-CD30-CAR-transduced T cells, beginning in the first stage with the aim of over 30% reaction rate among 15 patients with B cell malignancies. Only when the expected reaction rate is achieved the 30 patients left can be recruited.
  Interventions: Biological: Anti-CD30-CAR-transduced T cells

INTERVENTIONS:
Biological: Anti-CD30-CAR-transduced T cells — The first 3 enrolled patients will receive autologous-derived CD30-targeted CAR-T cells on day 1, 2 and 3 with respective 10%, 30% and 60% of the total expected dosage after receiving lymphodepleting chemotherapy. If the 3 patients don't display severe toxicity, the next patients enrolled will get infused in 2 days with respective 40% and 60% total dosage.
  Other Names: CD30-targeted CAR-T cells

SUMMARY:
The overall purpose of this study is to explore the therapeutic effect of BCMA-targeted chimeric antigen receptor T(CAR-T) cells in the treatment of lymphocyte derived malignancies.

DETAILED DESCRIPTION:
CD30 is originally described as a marker of Hodgkin's and Reed-Sternberg cells in Hodgkin's lymphoma. CD30 antibody has been applied to treat lymphocyte derived malignancies. To explore the potency of CD30 in CAR-T therapy, this trial is designed and conducted to test the safety and effect of CD30-targeted CAR-T.

ELIGIBILITY:
Inclusion Criteria:

1. CD30-expressing lymphocyte malignancy must be assured and must be relapsed or refractory disease. According to current traditional therapies, there must be no available alternative curative therapies and subjects must be either ineligible for allogeneic stem cell transplant (SCT), have refused SCT, or have disease activity that prohibits SCT at this time.
2. Patients enrolled must have an evaluated score above 60 with KPS.
3. CD30 expression of the malignant cells must be detected by immunohistochemistry or by flow cytometry. In general immunohistochemistry will be used for lymph node biopsies, flow cytometry will be used for peripheral blood and bone marrow samples.
4. Gender is not limited, age from 14 years to 75 years.
5. Patients must have measurable or evaluable disease at the time of enrollment, which may include any evidence of disease including minimal residual disease detected by flow cytometry, cytogenetics, or polymerase chain reaction (PCR) analysis.
6. Patients are expected to survive for more than 3 months by their physicians at the time of enrollment.
7. Adequate absolute CD3 count estimated need to be assured for obtaining target cell dose based on dosage cohorts.
8. Subjects with the following CNS status are eligible only in the absence of neurologic symptoms suggestive of CNS leukemia, such as cranial nerve palsy:

   CNS 1, defined as absence of blasts in cerebral spinal fluid (CSF) on cytospin preparation, regardless of the number of WBCs; CNS 2, defined as presence of < 5/uL WBCs in CSF and cytospin positive for blasts, or > 5/uL WBCs but negative by Steinherz/Bleyer algorithm CNS3 with marrow disease who has failed salvage systemic and intensive IT chemotherapy (and therefore not eligible for radiation)
9. Ability to give informed consent.
10. Cardiac function: Left ventricular ejection fraction greater than or equal to 40% by MUGA or cardiac MRI, or fractional shortening greater than or equal to 28% by ECHO or left ventricular ejection fraction greater than or equal to 50% by ECHO.
11. Renal function: Creatinine level of peripheral blood is required no greater than 133umol/L.
12. Females of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects on the fetus.
13. Patients with history of allogeneic stem cell transplantation are eligible if there is no evidence of active GVHD and no longer taking immunosuppressive agents for at least 30 days prior to enrollment.
14. Patients volunteer to participate in the research.

Exclusion Criteria:

1. Evident signs suggesting that patients are potentially allergic to cytokines.
2. Frequent infection history and recent infection is uncontrolled.
3. Patients with concomitant genetic syndrome: patients with Down syndrome, Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome
4. Active acute or chronic graft-versus-host disease (GVHD) or requirement of immunosuppressant medications for GVHD within 4 weeks of enrollment.
5. Concurrent use of systemic steroids or chronic use of immunosuppressant medications. Recent or current use of inhaled steroids is not exclusionary. For additional details regarding use of steroid and immunosuppressant medications.
6. Pregnancy and nursing females.
7. HIV infection.
8. Active hepatitis B or active hepatitis C.
9. Participation in a prior investigational study within 4 weeks prior to enrollment or longer if required by local regulation. Participation in non-therapeutic research studies is allowed.
10. Class III/IV cardiovascular disability according to the New York Heart Association Classification.
11. Patients with a known history or prior diagnosis of other serious immunologic, malignant or inflammatory disease.
12. Other situations researchers think not eligible for participation in the research.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Adverse Events That Are Related to Treatment | 3 years
  Determine the toxicity profile of the BCMA targeted CAR T cells with Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0.

SECONDARY OUTCOMES:
In vivo existence of Anti-CD30 CAR-T cells | 3 years
Reaction Rate of Treatment | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Qian, MD, PhD, Principal Investigator — Biotherapy Center of Southwest Hospital
Locations (1):
- Southwest Hospital of Third Millitary Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided